CLINICAL TRIAL: NCT05287893
Title: A Phase 1b Study to Characterise the Pharmacokinetic/Pharmacodynamic Relationship of Pyronaridine in Healthy Adult Participants Experimentally Infected With Blood Stage Plasmodium Falciparum.
Brief Title: Pyronaridine in Healthy Adult Participants Infected With Blood Stage Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: QIMR Berghofer Medical Research Institute (Other); Southern Star Research (Industry); Swiss BioQuant (Industry); Children's Health Queensland Hospital and Health Service (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MMV_Pyronaridine_21_01
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Malaria,Falciparum; Malaria; Malaria Recrudescence; Parasitemia; Protozoan Infections; Parasitic Disease
Keywords: Malaria; Malaria,Falciparum; Malaria Recrudescence; Parasitaemia; Pyronaridine
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Parasitemia; Protozoan Infections; Parasitic Diseases | interventions — pyronaridine

STUDY DESIGN:
Intervention Model Description: Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship. Each cohort will comprise up to three dose groups, with participants randomised to a dose group on the day of dosing. The highest dose of pyronaridine administered will be no more than 720 mg; the lowest dose administered will be no less than 180 mg. The proposed dosing regimen for the Cohort 1, assuming six participants are enrolled, is as below. If less than six participants are enrolled the Safety Data Review Team (SDRT) will meet between Day 0 and Day 8, to decide on the dose/s to be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pyronaridine 360 mg (Experimental): Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
  Interventions: Drug: Pyronaridine; Biological: P. falciparum IBSM infection
- Pyronaridine 540 mg (Experimental): Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
  Interventions: Drug: Pyronaridine; Biological: P. falciparum IBSM infection
- Pyronaridine 720 mg (Experimental): Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
  Interventions: Drug: Pyronaridine; Biological: P. falciparum IBSM infection
- Not treated (Other): This inoculated participant was treated with rescue medication instead of pyronaridine due to testing positive for SARS-CoV-2 (COVID-19).
  Ten (10) participants were inoculated with P. falciparum and were included in the Full Analysis Set (FAS). Nine (9) inoculated participants were subsequently administered pyronaridine, and were included in the IMP Set, PK Analysis Set, PD Analysis Set, and the PK/PD Analysis Set. Some of the 18S qPCR data for the inoculated participant who was not administered pyronaridine was used in the PD model for PK/PD analyses.
  Interventions: Biological: P. falciparum IBSM infection

INTERVENTIONS:
Drug: Pyronaridine — Single dose
  Arms: Pyronaridine 360 mg; Pyronaridine 540 mg; Pyronaridine 720 mg
Biological: P. falciparum IBSM infection — Induced Blood Stage Malaria

SUMMARY:
This is an open-label, adaptive study that will utilise the P. falciparum induced blood stage malaria (IBSM) model to characterise the pharmacokinetic/pharmacodynamic (PK/PD) profile of pyronaridine. Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. Following a screening period of up to 28 days, cohorts of up to 6 healthy participants will be enrolled. Each participant will be inoculated intravenously on Day 0 with P. falciparum infected erythrocytes. Participants will be followed up daily on Days 1 to 3, and will attend the clinical unit once on Days 4, 5, 6 and 7 for clinical evaluation and blood sampling. Participants will be admitted to the clinical trial unit on Day 8 for a single oral dose of pyronaridine.

Different doses of pyronaridine will be administered across and within cohorts. Participants will be randomised to a dose group on the day of dosing. The highest dose of pyronaridine administered will be no more than 720 mg; the lowest dose administered will be no less than 180 mg.

Each subsequent cohort will be composed of up to 3 dose groups. The Safety Data Review Team (SDRT) will review all available safety and tolerability data from the previous cohort/s prior to inoculation of the next cohort.

Participants will be confined in the clinical unit for at least 96 h (Days 8 - 12) to monitor the safety and tolerability of pyronaridine dosing. Upon discharge from the clinical unit participants will be monitored on an outpatient basis up to Day 50±2. Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2 or earlier.

DETAILED DESCRIPTION:
This is an open-label, adaptive study that will utilise the P. falciparum induced blood stage malaria (IBSM) model to characterise the pharmacokinetic/pharmacodynamic (PK/PD) profile of pyronaridine.

Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. Following a screening period of up to 28 days, cohorts of up to 6 healthy participants will be enrolled. Each participant will be inoculated intravenously on Day 0 with approximately 2,800 viable P. falciparum infected erythrocytes. Participants will be followed up daily via phone call or text message on Days 1 to 3 post-inoculation to solicit any adverse events. Participants will attend the clinical unit once on Days 4, 5, 6 and 7 for clinical evaluation and blood sampling to monitor the progression of parasitaemia, using quantitative polymerase chain reaction (qPCR) targeting the gene encoding 18S rRNA (referred to hereafter as malaria 18S qPCR). Participants will have a nasopharyngeal aspirate (NPA) for SARS-CoV-2 on Day 6 am in the event that there is community transmission in South East Queensland of SARS-CoV-2. Participants will also have blood collected on Day 7 am to monitor haematology and biochemistry. Participants will be admitted to the clinical trial unit on Day 8 for dosing with the investigational medicinal product (IMP; pyronaridine) when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL. Pyronaridine will be administered as a single oral dose. Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship. Each cohort will comprise up to three dose groups, with participants randomised to a dose group on the day of dosing. The highest dose of pyronaridine administered will be no more than 720 mg; the lowest dose administered will be no less than 180 mg. The proposed dosing regimen for the Cohort 1, assuming six participants are enrolled, is as below. If less than six participants are enrolled the Safety Data Review Team (SDRT) will meet between Day 0 and Day 8, to decide on the dose/s to be administered.

Dose group

1A (n=2) 360 mg

1B (n=2) 540 mg

1C (n=2) 720 mg

Each subsequent cohort will be composed of up to 3 dose groups. If more than one dose is tested in a given cohort, subjects will be randomised after inoculation day (Day 0) but prior to Day 8. The dose/s administered to Cohort 2 and Cohort 3 will be selected based on PK/PD and safety data from the preceding cohort/s. The SDRT will review all available safety and tolerability data and PK/PD analysis outcomes from the previous cohort/s prior to inoculation of the next cohort. The study will conclude when sufficient data have been obtained to define the PK/PD parameters for pyronaridine (the primary endpoint).

A maximum sample size of 18 participants administered pyronaridine is expected to be sufficient to achieve the primary endpoint.

Participants will be confined in the clinical unit for at least 96 h (Days 8 - 12) to monitor the safety and tolerability of pyronaridine dosing and to ensure adequate clinical response against P. falciparum. During confinement, regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration. If participants are clinically well at the end of the confinement period, they will be discharged and monitored on an outpatient basis up to Day 50±2.

Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2 or earlier.

ELIGIBILITY:
Inclusion Criteria:

Demography

1. Male or female (non-pregnant, non-lactating) aged 18 to 55 years inclusive who will be contactable and available for the duration of the trial and up to two weeks following the EOS visit.
2. Total body weight greater than or equal to 50 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive). BMI is an estimate of body weight adjusted for height. It is calculated by dividing the weight in kilograms by the square of the height in metres.

   Health status
3. Certified as healthy by a comprehensive clinical assessment (detailed medical history and full physical examination).
4. Vital signs at screening (measured after 5 min in the supine position):

   * Systolic blood pressure (SBP) - 90-140 mmHg,
   * Diastolic blood pressure (DBP) - 40-90 mmHg,
   * Heart rate (HR) 40-100 bpm.
5. At Screening and pre-inoculation with the malaria challenge agent: normal standard mean of triplicate 12-lead electrocardiogram (ECG) parameters after 5 minutes resting in supine position in the following ranges:

   1. QTcF ≤450 msec (male participants); QTcF ≤470 msec (female participants);
   2. QRS 50-120 msec
   3. PR interval ≤ 210 msec for both males and females, and
   4. Normal ECG tracing unless the PI or delegate considers an ECG tracing abnormality to be not clinically relevant.
6. Women of childbearing potential (WOCBP) who anticipate being sexually active with a male during the trial must agree to the use of a highly effective method of birth control (see below) combined with a barrier contraceptive from the screening visit until 100 days after the last dose of pyronaridine (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose pyronaridine) and have a negative result on urine pregnancy test performed before inoculation with the malaria challenge agent.

Note:

a. Highly effective birth control methods include: combined (oestrogen and progestogen containing) oral/intravaginal/transdermal/implantable hormonal contraception associated with inhibition of ovulation, progestogen-only oral/injectable/implantable hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, or sexual abstinence or same sex relationship.

b. Female participants who are abstinent (from penile-vaginal intercourse) must agree to start a double method if they start a sexual relationship with a male during the study. Female participants must not be planning in vitro fertilisation within the required contraception period.

7. Women of non-childbearing potential (WONCBP) are defined as:

1. Natural (spontaneous) post-menopausal defined as being amenorrhoeic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level (FSH) >25 IU/L (or at the local laboratory levels for post-menopause)
2. Premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months before screening (as determined by participant medical history) 8. Males who have, or may have, female sexual partners of child bearing potential during the course of the study must agree to use a double method of contraception including condom plus diaphragm, or condom plus intrauterine device, or condom plus stable oral/transdermal/injectable/implantable hormonal contraceptive by the female partner, from the time of informed consent through to 70 days (covering a spermatogenesis cycle) after pyronaridine administration. Abstinent males must agree to start a double method if they begin sexual relationship with a female during the study and up to 70 days after the last dose of pyronaridine. Males with female partners of child-bearing potential that are surgically sterile, or males who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception.

   Regulations 9. Completion of the written informed consent process prior to undertaking any trial-related procedure.

   10. Must be willing and able to communicate and participate in the whole trial. 11. Agreement to adhere to Lifestyle Considerations (see Section 5.3) throughout trial duration 12. Agreement to provide current contact details (two telephone numbers including a mobile number and a responsible adult as an emergency contact) and a relevant email address.

   Exclusion Criteria:
   * Individual who lives alone, OR, does not satisfy the following criteria: Participants who live alone may be included on a case-by-case basis, following discussion with the Principal Investigator. Participants who live alone must identify and provide contact details of a support person who is aware of the participant's participation in the study and is available to provide assistance if required (for example with contacting the participant in the event that study staff are unable to, or with transporting the participant to and from the study site if required).

     2. Known hypersensitivity to pyronaridine, artesunate or any of its derivatives, artemether, lumefantrine or other artemisinin derivatives, proguanil/atovaquone, primaquine, or 4-aminoquinolines.

     3. Haematology, biochemistry or urinalysis results at screening or at the eligibility visit that are outside of Sponsor-approved clinically acceptable laboratory ranges (appendix) or are considered clinically significant by the PI or their delegate.

     4. Participation in any investigational product trial within the 12 weeks preceding pyronaridine administration.

     5. Symptomatic postural hypotension at screening (confirmed on two consecutive readings), irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 min when changing from supine to standing position.

     6. Any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing, or other food or drug allergy that the Investigator considers may impact on participant safety. Participants with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic at the time of dosing can be enrolled in the trial.

     7. History of convulsion (including drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood (< 5 years) is not an exclusion criterion.

     8. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease, diabetes, progressive neurological disease, severe malnutrition, hepatic or renal disease. Acute or progressive hepatic or renal disease, porphyria, psoriasis, rheumatoid arthritis, asthma (excluding childhood asthma, or mild asthma with preventative asthma medication required less than monthly), or epilepsy.

     9. History of malignancy of any organ system (other than localised basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within five years of screening, regardless of whether there is evidence of local recurrence or metastases.

     10. Individuals with history of schizophrenia, bipolar disorder psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including generalised anxiety disorder.

     11. Individuals who have been hospitalised within five years prior to enrolment for either a psychiatric illness or due to danger to self or others.

   History of an episode of mild/moderate depression lasting more than 6 months that required pharmacological therapy and/or psychotherapy within the last 5 years; or any episode of major depression.

   The Beck Depression Inventory-II (BDI-II) will be used as a validated tool for the assessment of depression at screening. In addition to the conditions listed above, participants with a score of 20 or more on the BDI-II and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. These participants will be referred to a general practitioner or medical specialist as appropriate. Participants with a BDI-II score of 17 to 19 may be enrolled at the discretion of an Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the participant or to the execution of the trial and interpretation of the data gathered.

   13. History of recurrent headache (e.g. tension-type, cluster, or migraine) with a frequency of ≥2 episodes per month on average and severe enough to require medical therapy, during the 2 years preceding screening.

   14. Presence of clinically significant infectious disease or fever (e.g., sublingual temperature ≥38.5°C) within the five days prior to inoculation.

   15. Blood product donation to any blood bank during the 8 weeks (whole blood) or 4 weeks (plasma and platelets) prior to admission in the clinical unit on Day 8.

   16. History or presence of alcohol abuse (alcohol consumption more than 40 g/4 units/4 standard drinks per day), or drug habituation, or any prior intravenous usage of an illicit substance.

   17. Any individual who currently (within 14 days prior to inoculation) smokes >5 cigarettes/day.

   18. Breastfeeding or lactating; positive serum pregnancy test at screening, positive urine pregnancy test upon admission or at other time points as specified by schedule of activities tables.

   19. Any COVID-19 vaccine within 14 days of inoculation, any other vaccination within 28 days of IMP intake, and any vaccination (including COVID-19 initial or second dose) planned up to the final follow-up visit.

   20. Any corticosteroids, anti-inflammatory drugs (excluding commonly used over-the-counter anti-inflammatory drugs such as ibuprofen, acetylsalicylic acid, diclofenac), immunomodulators or anticoagulants within the past three months. Any individual currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration potentially associated with hypothalamic-pituitary-adrenal axis suppression within the past year.

   21. Use of prescription drugs (excluding contraceptives) or non-prescription drugs or herbal supplements (such as St John's Wort), within 14 days or five half-lives (whichever is longer) prior to inoculation. Limited use of other non-prescription medications or dietary supplements, not believed to affect participant safety or the overall results of the trial, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the PI. Participants are requested to refrain from taking non-approved concomitant medications from recruitment until the conclusion of the trial.

   22. Cardiac/QT risk: Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.

   History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.

   23. Any history of malaria or participation in a previous malaria challenge trial or malaria vaccine trial.

   24. Must not have had malaria exposure that is considered by the PI or their delegate to be significant. This includes but is not limited to: history of having travelled to or lived (>2 weeks) in a malaria-endemic region during the past 12 months or planned travel to a malaria-endemic region during the course of the trial; history of having lived for >1 year in a malaria-endemic region in the past 10 years; history of having ever lived in a malaria-endemic region for more than 10 years inclusive. For endemic regions see https://malariaatlas.org/explorer/#/, Bali is not considered a malaria-endemic region.

   25. Has evidence of increased cardiovascular disease risk (defined as >10%, 5-year risk for those greater than 35 years of age, as determined by the Australian Absolute Cardiovascular Disease Risk Calculator [http://www.cvdcheck.org.au/]). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, total and HDL cholesterol (mmol/L), and reported diabetes status.

   26. History of splenectomy. 27. Individual unwilling to defer blood donations to the Blood Service for at least twelve months after the EOS visit.

   28. Individual who has ever received a blood transfusion. 29. Any recent (<6 weeks) therapy with an antibiotic or drug with potential antimalarial activity (e.g. chloroquine, piperaquine phosphate, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, doxycycline etc.).

   General conditions 30. Any individual who, in the judgement of an Investigator, is likely to be non-compliant during the trial, or is unable to cooperate because of a language problem or poor mental development.

   31. Any individual in the exclusion period of a previous trial according to applicable regulations.

   32. Any individual who is an Investigator, research assistant, pharmacist, trial coordinator, or other staff thereof, directly involved in conducting the trial.

   33. Any individual without good peripheral venous access. Biological status 34. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).

   35. Positive urine drug test. Any drug listed in the urine drug screen unless there is an explanation acceptable to an Investigator (e.g., the participant has stated in advance that they consumed a prescription or over-the-counter product that contained the detected drug) and the participant has a negative urine drug screen on retest by the pathology laboratory.

   36. Severe G6PD deficiency. 37. Positive alcohol breath test. 38. Positive for SARS-CoV-2 by PCR. NPA testing is to occur between Day -3 to Day -1 but only in the event that there is community transmission in South East Queensland (see section 8.3.7) 39. Positive for red cell antibodies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Möhrle, PhD, Study Director — Medicines for Malaria Venture
Locations (2):
- Australia (2):
  - South Bank, Brisbane, Queensland
  - USC Clinical Trials, Morayfield, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant received the IBSM inoculum on Day 0 but tested positive for covid-19 before randomisation to an IMP dose on Day 8, and received the malaria rescue medication instead.
  Participants were randomised to 3 possible doses in cohort 1. Following a safety and PK/PD modelling data review of cohort 1 the number of participants to receive each dose in cohort 2 was determined.
  Upon cohort 1 and 2 safety and PK/PD data review the endpoint could be met and cohort 3 was not required.
Groups:
- Cohort 1: Pyronaridine 360 mg; Cohort 1: Pyronaridine 540 mg; Cohort 1: Pyronaridine 720 mg; Cohort 2: Pyronaridine 360 mg; Cohort 2: Pyronaridine 540 mg: Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL. Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship. Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
- Untreated: This inoculated participant was treated with rescue medication instead of pyronaridine due to testing positive for SARS-CoV-2 (COVID-19).
  Ten (10) participants were inoculated with P. falciparum and were included in the Full Analysis Set (FAS). Nine (9) inoculated participants were subsequently administered pyronaridine, and were included in the IMP Set, PK Analysis Set, PD Analysis Set, and the PK/PD Analysis Set. Some of the 18S qPCR data for the inoculated participant who was not administered pyronaridine was used in the PD model for PK/PD analyses.
Period: Initial Randomization and PKPD Modelling
Arm/Group | Cohort 1: Pyronaridine 360 mg | Cohort 1: Pyronaridine 540 mg | Cohort 1: Pyronaridine 720 mg | Untreated | Cohort 2: Pyronaridine 360 mg | Cohort 2: Pyronaridine 540 mg
Started | 2 | 2 | 1 | 1 | 0 (NA for period 1.) | 0 (NA for period 1.)
Completed | 2 | 2 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2 Dosing and Modelling
Arm/Group | Cohort 1: Pyronaridine 360 mg | Cohort 1: Pyronaridine 540 mg | Cohort 1: Pyronaridine 720 mg | Untreated | Cohort 2: Pyronaridine 360 mg | Cohort 2: Pyronaridine 540 mg
Started | 0 | 0 | 0 | 0 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 10 participants received inoculum and were included in the Full Analysis Set. 9 inoculated participants received 360mg (n=4), 560mg (n=4), or 720mg (n=1) pyronaridine, and included in the IMP Set, PK Analysis Set, PD Analysis Set, and the PK/PD Analysis Set. Some of the 18S qPCR data for the inoculated participant who was not administered pyronaridine was used in the PD model for PK/PD analyses.
  Analysis and results were grouped per dose/arm, not per cohort.
Groups:
- Pyronaridine 360 mg; Pyronaridine 540 mg; Pyronaridine 720 mg: Healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL. Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship. Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
- Total: Total of all reporting groups
Arm/Group | Pyronaridine 360 mg | Pyronaridine 540 mg | Pyronaridine 720 mg | Untreated | Total
Number analyzed (Participants) | 4 | 4 | 1 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.08 (7.46) | 36.0 (14.81) | 19.0 (NA) — n=1 | 42.0 (NA) — n=1 | 32.8 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 3
  Male | 4 | 3 | 0 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2 | 4 | 1 | 1 | 8
  Race: Asian | 1 | 0 | 0 | 0 | 1
  Race: Other | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 4 | 1 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Emax
Description: Maximum drug killing rate, calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data.
Time Frame: Day 8 to Day 50+/-2
Population: The PK analysis set will include all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study treatment and experienced no protocol deviations with relevant impact on PK data.
  Emax is calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan, so there is only 1 Emax result.
Measure: Mean (Standard Error); unit: Maximum clearance rate (1/hour)
Groups:
- IBSM Challenge and Pyronaridine PK/PD Population Profile: Ten (10) participants were inoculated with P. falciparum and were included in the Full Analysis Set (FAS). Inoculation occurred on Day 0 with participants receiving approximately 2,800 viable P. falciparum-infected erythrocytes intravenously.
  Day 8, nine (9) participants received pyronaridine when parasitaemia for the majority of participants was expected to be above 5,000 parasites/mL. Different doses of pyronaridine were administered across and within cohorts in order to effectively characterise the PK/PD relationship. Regular safety assessments were performed and blood collected to monitor parasite clearance and pyronaridine concentration. These 9 participants received compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier, and were included in the IMP Set, PK Analysis Set, PD Analysis Set, and the PK/PD Analysis Set. One (1) inoculated participant was treated with rescue medication instead of pyronaridine due to testing positive for SARS-CoV-2 (COVID-19). Some of the 18S qPCR data for the inoculated participant who was not administered pyronaridine was used in the PD model for PK/PD analyses.
Arm/Group | IBSM Challenge and Pyronaridine PK/PD Population Profile
Number analyzed (Participants) | 10
Maximum clearance rate (1/hour) | 0.201 (3.87)

2. Primary Outcome: EC50
Description: Half Maximal Effective Concentration Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data.
Time Frame: Day 8 to Day 50+/-2
Population: Full analysis set Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data.
Measure: Mean (Standard Error); unit: μg/mL
Arm/Group | IBSM Challenge and Pyronaridine PK/PD Population Profile
Number analyzed (Participants) | 10
μg/mL | 0.00575 (11.3)

3. Primary Outcome: Hill Coefficient
Description: Hill coefficient is the slope of the drug concentration-response curve (i.e. response in this study is the parasite killing). Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data.
  The "Emax-model" assumes a direct effect of concentrations on parasite killing/clearance, such as:
  Kill = Emax x (Cc^Hill /(Cc^Hill + EC50^Hill))
  where Cc is the concentration in the central compartment, Emax is the maximum effect of the drug, EC50 is the concentration that results in 50% of the maximum effect, and Hill is the Hill coefficient.
Time Frame: Day 8 to Day 50+/-2
Population: Full analysis set. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data
Measure: Mean (Standard Error); unit: Hill Coefficient
Arm/Group | IBSM Challenge and Pyronaridine PK/PD Population Profile
Number analyzed (Participants) | 10
Hill Coefficient | 6.62 (2.42)

4. Primary Outcome: Minimum Inhibitory Concentration (MIC)
Description: MIC is defined as the concentration when drug killing equals the parasite growth, i.e., the time at which the minimum parasite concentration is observed. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
Time Frame: Day 8 to Day 50+/-2
Population: Full analysis set. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IBSM Challenge and Pyronaridine PK/PD Population Profile
Number analyzed (Participants) | 10
ng/mL | 5.5 [4.3 to 6.9]

5. Primary Outcome: Minimal Parasiticidal Concentration (MPC90)
Description: MPC90 is defined as the concentration at which the clearance effect is at 90% of the maximum. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
Time Frame: Day 8 to Day 50+/-2
Population: as for outcome 4
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IBSM Challenge and Pyronaridine PK/PD Population Profile
Number analyzed (Participants) | 10
ng/mL | 8 [6.4 to 10]

6. Primary Outcome: Parasite Reduction Ratio in 48 h (log10PRR48)
Description: PRR48 is defined as the parasite reduction ratio achieved within 48 hours, usually given as the reduction of values on log10 transformed scale. PRR48 provides an efficacy estimate of anti-malarial treatment and is the ratio of the parasite density over a 48 hour time-period. PRR48 is estimated using the slope of the optimal fit of the log-linear relationship of the parasitemia decay. Optimal fit is derived using the geometric mean parasitemia data (i.e. 18S qPCR measuring all blood stage malaria parasites). Optimal fit of log-linear parasitemia by time relationship is determined using left and right censoring to systematically remove potential lag phase and tail phase of parasitemia decay.
  The PRR48 was calculated per subject in MMV_PYR using daily PCR data; and if the model fit was adequate for the subject (defined as overall model p-value<0.001), the slope and corresponding standard error (SE) from the log-linear regression was used to calculate the overall dose-specific PRR48
Time Frame: Day 8 to Day 50+/-2
Population: PK analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: log[(parasites/mL)/hour]
Groups:
- Pyronaridine 360 mg: Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with pyronaridine when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL. Different doses of pyronaridine will be administered across and within cohorts in order to effectively characterise the PK/PD relationship. Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and pyronaridine concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 47±2, or earlier.
  Pyronaridine: Single dose P. falciparum IBSM infection: Induced Blood Stage Malaria
Arm/Group | Pyronaridine 360 mg | Pyronaridine 540 mg | Pyronaridine 720 mg
Number analyzed (Participants) | 4 | 4 | 1
log[(parasites/mL)/hour] | 2.58 [2.43 to 2.74] | 2.53 [2.37 to 2.68] | 2.85 [2.65 to 3.06]

ADVERSE EVENTS:
Time Frame: The period of observation for collection of AEs extends from the time of inoculation with the malaria challenge agent (Day 0) to EOS (Day 50+/-2). A total maximum of 53 days.
Arm/Group | Pyronaridine 360 mg | Pyronaridine 540 mg | Pyronaridine 720 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine 360 mg (N=4) | Pyronaridine 540 mg (N=4) | Pyronaridine 720 mg (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Administration site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (3) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (3) | 3 (4) | 1 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (3) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 1 (4) | 3 (4) | 1 (5)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (17) | 2 (12) | 1 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI's organisation will prepare the manuscript once the Clinical Study Report finalisation (within 12 months of trial completion). The Sponsor organisation will have 45 days to review prior to submission for for publication.

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT05287893/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT05287893/SAP_001.pdf